CLINICAL TRIAL: NCT05760144
Title: Endometrial Biopsy in Progestin Contraceptive Users
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alison Edelman, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 25084
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-08

CONDITIONS: Contraception
MeSH Terms: interventions — N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DMPA (Active Comparator)
  Interventions: Drug: DMPA
- Etonogestrel implant (Active Comparator)
  Interventions: Drug: Etonogestrel implant

INTERVENTIONS:
Drug: DMPA — The participant will receive the contraceptive injectable, Depo-Provera at the enrollment visit and at 3, 6, 9, and 12 months. Participants will have endometrial biopsies at the enrollment visits and at 3, 6, and 12 months.
  Other Names: Depo-Provera
  Arms: DMPA
Drug: Etonogestrel implant — The participant will receive the contraceptive implant, Nexplanon at the enrollment visits and have endometrial biopsies at the enrollment visits and at 3, 6, and 12 months.
  Other Names: Nexplanon
  Arms: Etonogestrel implant

SUMMARY:
The purpose of the study is to learn more about menstrual changes in progestin contraception users. The investigators are hoping to find out what changes in the endometrium lead to different bleeding patterns during the first year of progestin contraception use. Participants will choose to receive the contraceptive implant (Etonogestrel implant also called Nexplanon) or the contraceptive injectable (Depo-medroxyprogesterone acetate (DMPA) also called Depo-Provera) for up to 12 months. They will be asked to have 4 endometrial biopsies over the course of the study, as well as blood draws, physical exams, and pregnancy tests. Participants will also use a daily text message or email diary to report bleeding patterns. This study's plan is to comprehensively phenotype bleeding patterns and profile the entire endometrium using single-cell RNA seq data (sCRNAseq).

ELIGIBILITY:
Inclusion Criteria:

* 18-4 0 years of age at time of enrollment in good general health
* Regular menstrual cycles (25-35 day cycle length with bleeding 8 days or less)
* Body Mass Index of 19-35
* Confirmed ovulation with a screening serum progesterone of greater than 3ng/mL
* No contraindications to DMPA or hormonal implant

Exclusion Criteria:

* Hormonal or intrauterine contraceptives or other hormone use prior to start of study enrollment [No oral hormonal contraceptives or other hormones for at least one month, no implantable contraceptives or hormonal or non-hormonal intrauterine device for at least two months (2 cycles), no injectable hormonal contraceptives or other hormones in past 9 months from the most recent injection and resumption of regular menstrual cycles]. Of note, patients could have used an implant or DMPA in past but must have the same washout time periods as noted before.
* Any known uterine pathology (endometriosis, leiomyoma or adenomyosis; bacterial, fungal or viral infection, active cervicitis). For bacterial infection such as gonorrhea (GC) /chlamydia (CT) enrollment should be delayed until treatment complete. For vaginitis (bacterial vaginosis or yeast) enrollment can occur at time of diagnosis if patient prefers. Test of cure is not required to proceed with enrollment.
* Positive gonorrhea/chlamydia screening performed at screening visit, unless treated as noted above.
* Routine or chronic use of non-steroidal anti-inflammatory drugs (NSAIDs once daily or more 14 or more days per month)
* Abnormal uterine bleeding
* Polycystic ovary syndrome
* Currently pregnant or planning pregnancy during the study
* Less than 6 month postpartum or breastfeeding, post abortion 6 weeks, not breast/chest feeding (cessation 4-6 weeks from enrollment)
* Centers for Disease Control Medical Eligibility for Contraceptive use category 3 or 4 for contraceptive usage (Current or prior medical history of thrombosis or thromboembolic disorders, Liver tumors or active liver disease, Current or prior medical history of breast cancer, Hypertension defined as 160/100 or greater, Ischemic heart disease or multiple risk factors for atherosclerotic cardiovascular disease, Rheumatoid arthritis on immunosuppressive therapy, History of stroke, Systemic lupus erythematosus, Unexplained vaginal bleeding, Diabetes of greater than 20 years duration or with evidence with end-organ disease)
* Anticoagulation use
* Bleeding dyscrasia
* Use of P450 pathway inducing drug(s)
* Inability to tolerate uterine sounding (at screening visit)
* Chronic use of Cannabidiol, THC, or marijuana (More than 3 times per week). Of note, patients could have used Cannabidiol, THC, or marijuana chronically in past, but must have a washout time period of no use for at least one month prior to the study.
* Chronic use of cigarettes (More than 1 cigarette per week). Of note, patients could have used cigarettes chronically in past, but must have a washout time period of no use for at least six months prior to the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who experienced endometrial changes | Baseline to 6 months
  The proportion of participants who experienced endometrial changes, as defined by any changes in gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States